CLINICAL TRIAL: NCT03359408
Title: Supporting Elderly People With Cognitive Impairment During and After Hospital Stays- Intersectoral Care Management [Verbundprojekt Intersec-CM - sektorenübergreifendes Care Management Zur Unterstützung Kognitiv beeinträchtigter Menschen während Und Nach Einem Krankenhausaufenthalt]
Brief Title: Supporting Elderly People With Cognitive Impairment During and After Hospital Stays- Intersectoral Care Management
Acronym: intersec-CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Medicine Greifswald (Other); Evangelisches Klinikum Bethel gGmbH (Unknown); Jena University Hospital (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, René Thyrian, Working Group leader, German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR007
Record Dates: First submitted 2017-11-16; First posted 2017-12-02 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Dementia; Cognitive Impairment; Neurodegenerative Diseases
Keywords: Health care; Dementia care; Collaborative care; Discharge management; Hospital; Primary care
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): Care as usual, no intervention, just observation of natural change/ trajectories over time
- Dementia Care Management (DCM) (Experimental): Subjects in this arm will be provided with "Dementia Care Management" adapted to the intersectoral setting.
  Interventions: Behavioral: Dementia Care Management (DCM)

INTERVENTIONS:
Behavioral: Dementia Care Management (DCM) — A specialised discharge management, based on "Dementia Care Management" (DCM; Thyrian et al. 2017, Eichler, Thyrian, Fredrich et al. 2014, Eichler, Thyrian, Dreier et al. 2014, Dreier et al. 2016, ) will be applied to subjects with cognitive impairment. Specifically qualified will conduct comprehensive data assessments during the hospital stay, assess recommendations at discharge and assess unmet needs at home. Supported by a a computerized Intervention Management (IMS) and in close cooperation with the discharging hospital, treating physicians and other care providers, they will develop, implement and monitor a treatment and care plan. Interventional home visits will take place at the participants homes.
  Arms: Dementia Care Management (DCM)

SUMMARY:
Sectorisation of the German health care system causes inefficient treatment, especially in elderly with cognitive impairments. At time of transition from hospitals into primary care it lacks, among others, coordination of post-operative care or timely communication between healthcare providers. This results in deterioration of disease and comorbidities, higher rates of re-admission and institutionalizations. Models of collaborative care have shown their efficacy in primary care. Main goal is to test the effectiveness of Dementia Care Management (DCM) for people with cognitive impairment to improve treatment and care across the in-hospital and primary care sector.

The study design is a complex, longitudinal, multisite randomized controlled trial. It was designed to treat a hospital-based epidemiological cohort of people above the age of 70 with an adaption of DCM, a treatment proven to be effective in primary care, to the discharge setting. As part of this, specifically trained study staff will develop, implement and monitor a treatment and care plan, based on comprehensive assessments during the hospital stay, recommendations at discharge and unmet needs at home. For the 3 months after discharge study staff will coordinate treatment and care in close cooperation with the discharging hospital, treating physician and other care providers.

Expected results from the study should facilitate the implementation of intersectoral care management systematically on a large scale. Thus, the benefits shown in the trial would be available to a larger population. Results will not be limited to PCI, but rather to any people transitioning between the in-hospital and the primary care sector. Thus, the benefits would be available to elderly people in general.

DETAILED DESCRIPTION:
The German health care system is sectorized with health service providers offering a) outpatient treatment and care, b) inpatient treatment and care or c) rehabilitation. While treatment and care within these sectors can be considered to be of high quality, there is a lack of widely available approaches to deliver treatment and care across sectors. Treatment paths for people with chronic diseases or the requirements of elderly people suffering from multimorbidity need frequent transitions between sectors. However, in Germany boundaries of sectors are considered rigid and transitions between sectors are a threat to treatment continuity, which results in inefficient treatment. As this problem has been identified and described by the Advisory Council on the Assessment of Developments in the Health Care System (Sachverständigenrat zur Begutachtung der Entwicklung im Gesundheitswesen) already in 20121, different approaches have been proposed. This study addresses the lack of integrated cross-sectoral approaches to overcome the challenges caused by the sectorized German health care system.There is sound scientific evidence internationally and nationally that collaborative concepts of care can improve treatment and care of people with dementia in primary care (Thyrian et al. 2017). Those concepts are person-centered in the sense of a) taking into account the individual needs, circumstances and priorities, and b) aiming at outcomes relevant to the individuals life, like everyday functionality, (health related) quality of life and social inclusion.

The trial is a complex, longitudinal, multisite randomized controlled trial (intervention vs. care as usual). Recruitment of the study population will be conducted in two participating hospitals. After meeting the eligibility criteria, participants will be asked for written informed consent. With all participants a basic baseline assessment will be conducted (T0) in the hospital. After that they will be randomized in either the intervention group or control group. The intervention group will then receive the intervention, the control group care as usual. Further data assessments will be conducted at all participants´ home 3 months after discharge (T1) and at the participants´ home 12 months after discharge (T2). A process evaluation will also be applied in this study. Data assessment will be conducted by specifically trained study staff. Places of assessment are chosen for the highest possible convenience for the participants. Data assessments will include a) primary data from the participants being assessed, computer-assisted, face-to face and paper-pencil, b) secondary data from patient records in the hospital and from treating physicians.

The main research question of this protocol addresses the effectiveness of Dementia Care Management (DCM) in the intersectoral setting for people with cognitive impairment (PCI) in treatment and care across the in-hospital and primary care sector. The investigators will test the hypothesis if PCI receiving DCM initiated in hospitals and continued after discharge into ambulatory care do have better health and social outcomes after one year than PCI not receiving DCM. The patient-oriented minor hypotheses of this protocol are: ICM improves (a) health related quality of life sustainable, (b) social functioning and integration and (c) adequate treatment and care for dementia and co-morbidities in the ambulatory setting. It reduces (d) the risk for drug related problems in cognitive impairment and comorbidities and (e) the risk for re-admission to the hospital. The intervention prevents (f) incident delirium - given better awareness in respect to precipitating factors. The healthcare provider-oriented minor hypotheses are: ICM (a) reduces re-admission rates and thus saves costs in the inpatient setting. It increases (b) the chances to delay institutionalization significantly and thus saves costs from perspective of statutory health insurance. It (c) improves communication and exchange between treatment and care provider from different health care sectors sustainable. Furthermore, this protocol evaluates the process of implementing ICM along the main research question: How is ICM evaluated and rated among the different groups affected by it? Specific research questions are: What are the perceived benefits for (a) the providers (in the inpatient setting, (b) providers in the ambulatory setting, (c) the PCI and their caregiver? Is ICM evaluated as (d) improving communication and exchange between treatment and care provider from different health care sectors sustainable? And last not least, (e) what are the enablers and barriers to implement ICM in routine care?

ELIGIBILITY:
Inclusion Criteria:

* 70+ years
* minimum hospital stay of 5 days
* living at home
* positive cognitive screening (MMSE)
* written informed consent

Exclusion Criteria:

* stroke

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 401 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Instrumental and Physical Functionality | Assessed at T0 (time of hospital admission), at T1 (3 months after discharge) and T2 (12 months after discharge)
  The Bayer Activities of Daily Living Scale (B-ADL; Erzigkeit et al., 2001) will be used. It consists of 25 items indicating everyday problems/ challenges. Their occurence is rated on a scale of 1 "never", to 10 "always". All ratings are added and divided by the number of items. This yields a mean score of 1 to 10, where 1 indicates the lowest possible impairment and 10 indicates the highest possible impairment.
Re-Admission to Hospital | Assessed 3 months and 12 months after the time of hospital discharge (T1, T2).
  Participant will be asked if he/she has been hospitalized within the last 12 months. This is one item in the "the Questionnaire for the Use of Medical and Non-Medical Services in Old Age"; FIMA; (Seidl et al., 2015) which is administered to assess utilisation of health services.
Institutionalisation | Assessed 12 months after the time of hospital discharge (T2).
  Participant will be asked if he/she changed his/her living situation during the last 12 months. The answer will be validated with the question what the participants current living situation is. Both questions are items in the "the Questionnaire for the Use of Medical and Non-Medical Services in Old Age"; FIMA; (Seidl et al., 2015) which is administered to assess utilisation of health services.

SECONDARY OUTCOMES:
Change in Quality of Life | Assessed at T1 (time of hospital discharge, on average 12 days after admission), T2 (3 months after T1) and T3 (12 months after T1)
  Quality of life will be assessed using the EQ-5D, a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. As proxy rating the questionnaire QUALIDEM [Ettema et al., 2007] will be used to assess the quality of life of people with dementia aged ≥ 65 years.
Frailty | Assessed at T0 (time of hospital admission), at T1 (3 months after discharge) and T2 (12 months after discharge)
  Frailty will be assessed using the Edmonton frailty scale (EFS; Rolfson et al. 2006) will be used. The EFS is reliable tool in geriatric medicine to assess the frailty of older patients on the domains Cognition, General health status, Functional independence, Social support, Medication use, Nutrition, Mood, Continence and Functional performance.
Cognitive Status | Assessed at T0 (time of hospital admission), at T1 (3 months after discharge) and T2 (12 months after discharge)
  The Mini Mental State Examination (MMSE; Cockrell & Folstein, 1988) will be used. The MMSE is a 30-point questionnaire to measure cognitive impairment. The questions are grouped into seven categories, each representing a different cognitive domain or function: Orientation to time (5 points); Orientation to place (5 points); Registration of three words (3 points); Attention and Calculation (5 points); Recall of three words (3 points); Language (8 points) and Visual Construction (1 point). Scores of 25-30 out of 30 are considered normal; 21-24 as mild, 10-20 as moderate and <10 as severe impairment.
Resource Utilisation | Assessed at T1 (3 months after discharge) and T2 (12 months after discharge)
  The Resource Utilization in Dementia questionaire (RUD; Wimo et al., 2010) will be used to measure the frequency of utilisation of general physicians and physicians of other specialties, out-patient treatments, in-patient treatments, hospitalisations, institutionalisation and therapeutic appliances.
Use of Medical and Non-Medical Services | Assessed at T1 (3 months after discharge) and T2 (12 months after discharge)
  The Questionnaire for the Use of Medical and Non-Medical Services in Old Age [Fragebogen zur Inanspruchnahme medizinischer und nicht-medizinischer Versorgungsleistungen im Alter"; FIMA; Seidl et al., 2015) will be used. The FIMA examines socio-economic variables and other medical factors by determining health-related costs.
Behavioral and Psychological Symptoms of Dementia | Assessed at T0 (time of hospital admission), at T1 (3 months after discharge) and T2 (12 months after discharge)
  Neuropsychiatric Inventory (NPI; Cummings 1997) will be used. The NPI represents an interview by proxy on twelve dimensions of neuropsychiatric behaviors, i.e. delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The presence (0= no, 1= yes) is asked. If present, the severity (rated 1 through 3; mild to severe) and frequency (1 to 4, rarely to very often) of each neuropsychiatric symptom are rated on. Thus the score for each dimension ranges from 0 = not present, 1= mildly and rarely to 12 = severe and often. A total NPI score is calculated as the sum of the frequency by severity scores of each domain range: 0 to 144, the higher the more neuropsychiatric symptomatic).
Depression | Assessed at T1 (3 months after discharge) and T2 (12 months after discharge)
  The short form of the Geriatric Depression Scale (GDS; Yesavage & Sheikh,1986) will be used. It consists of 15 questions. One point is conferred for each positively answered question. Scores of 11 - 15 indicate the presence of depression, 5 - 10 a mild depression and 0 - 5 no depression.
Caregiver Burden | Assessed at T1 (time of hospital discharge, on average 12 days after admission), T2 (3 months after T1) and T3 (12 months after T1)
  The revised version of the Zarit-Burden Inventory (ZBI; Zarit et al., 1980) will be used.The revised version ZBI is a caregiver self-report measure to examine burden which is associated with functional/behavioural impairments and home care situation. It contains 22 items using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).Total scores range from 0 indicating low burden to 88 indicating high burden.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen René Thyrian, PhD, Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (4):
- Germany (4):
  - University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Evangelisches Klinikum Bethel gGmbH, Bielefeld, North Rhine-Westphalia
  - Ruhr University Bochum (RUB), Bochum, North-Rhine-Westfalia
  - German Center for Neurodegenerative Diseases (DZNE), Greifswald

IPD SHARING:
Plan to Share IPD: Undecided
At the current status of the study, this has not been discussed with the funder and the research partners (11/13/17).

REFERENCES:
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Erzigkeit H, Lehfeld H, Pena-Casanova J, Bieber F, Yekrangi-Hartmann C, Rupp M, Rappard F, Arnold K, Hindmarch I. The Bayer-Activities of Daily Living Scale (B-ADL): results from a validation study in three European countries. Dement Geriatr Cogn Disord. 2001 Sep-Oct;12(5):348-58. doi: 10.1159/000051280. PMID 11455136
- [Background] Cockrell JR, Folstein MF. Mini-Mental State Examination (MMSE). Psychopharmacol Bull. 1988;24(4):689-92. No abstract available. PMID 3249771
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Zaudig M, Mittelhammer J, Hiller W, Pauls A, Thora C, Morinigo A, Mombour W. SIDAM--A structured interview for the diagnosis of dementia of the Alzheimer type, multi-infarct dementia and dementias of other aetiology according to ICD-10 and DSM-III-R. Psychol Med. 1991 Feb;21(1):225-36. doi: 10.1017/s0033291700014811. PMID 2047500
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Sheikh JI, Yesavage JA, Brooks JO 3rd, Friedman L, Gratzinger P, Hill RD, Zadeik A, Crook T. Proposed factor structure of the Geriatric Depression Scale. Int Psychogeriatr. 1991 Spring;3(1):23-8. doi: 10.1017/s1041610291000480. PMID 1863703
- [Background] Seidl H, Bowles D, Bock JO, Brettschneider C, Greiner W, Konig HH, Holle R. [FIMA--questionnaire for health-related resource use in an elderly population: development and pilot study]. Gesundheitswesen. 2015 Jan;77(1):46-52. doi: 10.1055/s-0034-1372618. Epub 2014 May 7. German. PMID 24806594
- [Background] Wimo A, Jonsson L, Zbrozek A. The Resource Utilization in Dementia (RUD) instrument is valid for assessing informal care time in community-living patients with dementia. J Nutr Health Aging. 2010 Oct;14(8):685-90. doi: 10.1007/s12603-010-0316-2. PMID 20922346
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Thyrian JR, Hertel J, Wucherer D, Eichler T, Michalowsky B, Dreier-Wolfgramm A, Zwingmann I, Kilimann I, Teipel S, Hoffmann W. Effectiveness and Safety of Dementia Care Management in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Oct 1;74(10):996-1004. doi: 10.1001/jamapsychiatry.2017.2124. PMID 28746708
- [Background] Thyrian JR. [People with dementia in primary care : Prevalence, incidence, risk factors and interventions]. Z Gerontol Geriatr. 2017 May;50(Suppl 2):32-38. doi: 10.1007/s00391-017-1223-5. Epub 2017 Apr 6. German. PMID 28386806
- [Background] Dreier A, Thyrian JR, Eichler T, Hoffmann W. Qualifications for nurses for the care of patients with dementia and support to their caregivers: A pilot evaluation of the dementia care management curriculum. Nurse Educ Today. 2016 Jan;36:310-7. doi: 10.1016/j.nedt.2015.07.024. Epub 2015 Jul 31. PMID 26277428
- [Background] Eichler T, Thyrian JR, Fredrich D, Kohler L, Wucherer D, Michalowsky B, Dreier A, Hoffmann W. The benefits of implementing a computerized intervention-management-system (IMS) on delivering integrated dementia care in the primary care setting. Int Psychogeriatr. 2014 Aug;26(8):1377-85. doi: 10.1017/S1041610214000830. Epub 2014 May 9. PMID 24811145
- [Background] Eichler T, Thyrian JR, Dreier A, Wucherer D, Kohler L, Fiss T, Bowing G, Michalowsky B, Hoffmann W. Dementia care management: going new ways in ambulant dementia care within a GP-based randomized controlled intervention trial. Int Psychogeriatr. 2014 Feb;26(2):247-56. doi: 10.1017/S1041610213001786. Epub 2013 Oct 23. PMID 24152974
- [Background] Thyrian JR, Fiss T, Dreier A, Bowing G, Angelow A, Lueke S, Teipel S, Flessa S, Grabe HJ, Freyberger HJ, Hoffmann W. Life- and person-centred help in Mecklenburg-Western Pomerania, Germany (DelpHi): study protocol for a randomised controlled trial. Trials. 2012 May 10;13:56. doi: 10.1186/1745-6215-13-56. PMID 22575023
- [Background] Rolfson DB, Majumdar SR, Tsuyuki RT, Tahir A, Rockwood K. Validity and reliability of the Edmonton Frail Scale. Age Ageing. 2006 Sep;35(5):526-9. doi: 10.1093/ageing/afl041. Epub 2006 Jun 6. No abstract available. PMID 16757522
- [Background] Ettema TP, Droes RM, de Lange J, Mellenbergh GJ, Ribbe MW. QUALIDEM: development and evaluation of a dementia specific quality of life instrument. Scalability, reliability and internal structure. Int J Geriatr Psychiatry. 2007 Jun;22(6):549-56. doi: 10.1002/gps.1713. PMID 17152121
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Derived] Boekholt M, Nikelski A, Schumacher-Schoenert F, Kracht F, Vollmar HC, Hoffmann W, Kreisel SH, Thyrian JR. Supporting older people with cognitive impairment during and after hospital stays with intersectoral care management (intersec-CM)-results of a randomised clinical trial. Age Ageing. 2025 Feb 2;54(2):afaf011. doi: 10.1093/ageing/afaf011. PMID 39912589
- [Derived] Kracht F, Boekholt M, Schumacher-Schonert F, Nikelski A, Chikhradze N, Lucker P, Vollmar HC, Hoffmann W, Kreisel SH, Thyrian JR. Describing people with cognitive impairment and their complex treatment needs during routine care in the hospital - cross-sectional results of the intersec-CM study. BMC Geriatr. 2021 Jul 12;21(1):425. doi: 10.1186/s12877-021-02298-4. PMID 34253180
- [Derived] Dehl T, Sauerbrey U, Dreier-Wolfgramm A, Nikelski A, Chikhradze N, Keller A, Laufer J, Schumacher-Schoenert F, Kreisel S, Thyrian JR, Hoffmann W, Vollmar HC. Intersectoral care management for older people with cognitive impairment during and after hospital stays [intersec-CM]: study protocol for a process evaluation within a randomised controlled trial. Trials. 2021 Jan 21;22(1):72. doi: 10.1186/s13063-021-05021-1. PMID 33478583
- [Derived] Nikelski A, Keller A, Schumacher-Schonert F, Dehl T, Laufer J, Sauerbrey U, Wucherer D, Dreier-Wolfgramm A, Michalowsky B, Zwingmann I, Vollmar HC, Hoffmann W, Kreisel SH, Thyrian JR. Supporting elderly people with cognitive impairment during and after hospital stays with intersectoral care management: study protocol for a randomized controlled trial. Trials. 2019 Aug 30;20(1):543. doi: 10.1186/s13063-019-3636-5. PMID 31470912